CLINICAL TRIAL: NCT05334849
Title: Prospectively Predict the Efficacy of Precise Immunotherapy Response of Gastric Cancer Based on Circulating Exosomal LncRNA-GC1 Biopsy
Brief Title: Prospectively Predict the Immunotherapy Response of Gastric Cancer Based on Circulating Exosomal LncRNA-GC1 Biopsy
Status: Completed | Type: Observational
Sponsor: Lin Chen (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, Director of Department of General Surgery, Chinese PLA General Hospital, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: irBiomarker
Record Dates: First submitted 2022-04-06; First posted 2022-04-19 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Advanced Gastric Carcinoma; Immunotherapy
Keywords: Circulating exosomal lncRNA-GC1; Advanced Gastric Carcinoma; Immunotherapy response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Circulating exosomal lncRNA-GC1 detection — Collect peripheral blood sample of 80 gastric cancer patients pre-treatment. Blood samples will be transferred to central lab to detect circulating exosomal lncRNA-GC1. Tumor response evaluation will be performed after two cycles of immunotherapy by CT/MRI based on RECIST.
  Clinical data, including tumor stage, metastastic organ, regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
To vertify the function of circulating exosomal lncRNA-GC1 on predicting and monitoring immunotherapeutic outcomes of GC

DETAILED DESCRIPTION:
The investigator's previous work identified circulating exosomal lncRNA-GC1 as a GC-specific tumor burden marker and this novel biomarker showed promising efficiency in monitoring disease progression during treatment.

Hence in this stuty, the investigator plan to recruit a prospective cohort to support the conclusions, and provide biomarkers to realize predicting and monitoring immunotherapeutic outcomes of GC.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Measurable disease according to the RECIST criteria
* Life expectancy of ≥3 month
* No prior chemotherapy of the study more than 4 weeks
* Immunotherapy regimens were included in the treatment

Exclusion Criteria:

* Other previous malignancy within 5 year
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study
* Pregnancy or lactation period
* Legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years and older
Study Population: All patients in this study were enrolled by the Department of General Surgery, Chinese PLA General Hospital for conventional therapy or clinical trials
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Levels of circulating exosomal lncRNA-GC1 | Circulating exosomal lncRNA-GC1 was detected, analysis and reported at the baseline
  Circulating exosomal lncRNA-GC1 was detected by the RT-PCR followed by isolating exosomes.
Levels of circulating exosomal lncRNA-GC1 | Circulating exosomal lncRNA-GC1 was detected, analysis and reported through study completion, average 1 year
  Circulating exosomal lncRNA-GC1 was detected by the RT-PCR followed by isolating exosomes.

SECONDARY OUTCOMES:
Survival outcomes of circulating exosomal lncRNA-GC1 | up to 3 years
  Analysis participants' survival with different levels of circulating exosomal lncRNA-GC1 detected by RT-PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided